CLINICAL TRIAL: NCT02818179
Title: Monitoring HDR Brachytherapy for Cervical Cancer by Optic and Thermal Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Tatiana Rabin MD, Senior Medical Doctor, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SHEBA-16-3171-RT-CTIL
Record Dates: First submitted 2016-06-16; First posted 2016-06-29 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: MALIGNANCY
MeSH Terms: conditions — Neoplasms | interventions — Thermography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing radiation (Other): In this study, patients undergoing radiation treatment will undergo thermography imaging during radiation treatment course. Patients will be evaluated with thermography imaging every week during the brachytherapy treatment for 5 procedures
  Interventions: Radiation: THERMOGRAPHY IMAGING

INTERVENTIONS:
Radiation: THERMOGRAPHY IMAGING

SUMMARY:
This research aims to investigate the correlation between tumor temperature difference and biological factors, such as size, metabolism, treatment response, and tumor aggressiveness.

In addition, normal tissue response to radiation therapy in treated organ will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* biopsy proven cervical cancer which will undergo definitive radiation

Exclusion Criteria:

* not eligible to sign informed consent

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The change in Infra-Red radiation emitted at wavelengths 0.8-1nm | Baseline and 4 weeks
  Measurement of IR

SECONDARY OUTCOMES:
Evaluating of efficacy of the radiation | 3 months after the treatment
  The thermal and the optic imaging will be taken and analyzed in order to evaluate the changing in the temperature of the cervix comparing to the baseline as the indication of the response to the radiotherapy